CLINICAL TRIAL: NCT02923700
Title: Leukocyte-rich PRP vs Leukocyte-poor PRP for the Treatment of Knee Cartilage Degeneration: a Randomized Controlled Trial
Acronym: PRP014
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRP014
Record Dates: First submitted 2016-09-30; First posted 2016-10-04 (Estimated); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Osteoarthritis
Keywords: platelet rich plasma; intra-articular injection; leukocytes
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Leukocyte-rich PRP group (Experimental): Three weekly knee intra-articular injections of leukocyte-rich PRP
  Interventions: Biological: Leukocyte-rich PRP intra-articular injections
- Leukocyte-poor PRP group (Experimental): Three weekly knee intra-articular injections of leukocyte-poor PRP
  Interventions: Biological: Leukocyte-poor PRP intra-articular injections

INTERVENTIONS:
Biological: Leukocyte-rich PRP intra-articular injections
  Arms: Leukocyte-rich PRP group
Biological: Leukocyte-poor PRP intra-articular injections
  Arms: Leukocyte-poor PRP group

SUMMARY:
Platelet-rich Plasma (PRP) is the most exploited biologic agents currently used for the treatment of osteoarthritis (OA) of different joints, in particular knee OA.

In previous studies, it has been showed its potential to reduce pain and improve functional status in patients treated by simple intra-articular injections. However, there are several PRP formulation currently available in clinical use, and therefore it is very difficult to compare data coming from trials using different products. The most debated aspect concerning PRP formulation is the role of leukocytes, which might stimulate an early inflammatory response in the joint due to the release of metalloproteases and other pro-inflammatory cytokines.

The investigators hypothesized that the presence of leukocytes in PRP could be clinically relevant in terms of outcome, so the present double blind randomized controlled trial was designed to compare leukocyte-rich and leukocyte-poor PRP injections for the treatment of knee OA.

A power analysis has been performed for the primary endpoint of IKDC (International Knee Documentation Committee) subjective score improvement at the 12-month follow-up for PRP. From a pilot study, a standard deviation of 15.2 points was found. With an alpha error of 0.05, a beta error of 0.2 and a minimal clinically significant difference of 6.7 points corresponding at 1/3 of the documented mean improvement, the minimum sample size was 83 for each group. Considering a possible drop out of 15%, 96 patients per group are required for total 192 patients, selected according to well-defined inclusion criteria (see 'Eligibility criteria' section). Patients are then assigned to two different treatment groups, according to a randomization list. The first group of treatment consists of three weekly intra-articular injections of autologous leukocyte-rich PRP, whereas the second group of patients will be treated by three intra-articular injections of leukocyte-poor PRP.

PRP will be obtained with the following procedure: a 300-ml autologous venous blood sample will undergo 2 centrifugations (the first at 1480 rpm for 6 minutes to separate erythrocytes, and a second at 3400 rpm for 15 minutes to concentrate platelets) to produced 20 ml of leukocyte-rich PRP. In case of patients allocated to receive leukocyte-poor PRP, a special filter will be then used to separate leukocytes and obtain leukocyte-poor PRP.

The total amount of PRP will be divided into 4 small units of 5 ml each. One unit is sent to the laboratory for analysis of platelet concentration and for a quality test, 3 units are stored at -30° C.

One week after the PRP production, the injective treatment starts, with 3 weekly injections. At the moment of the injection the syringe is properly covered to prevent the patient from discovering the substance he was receiving. After the injection, patients are sent home with instructions to limit the use of the leg for at least 24 h and to use cold therapy/ice on the affected area to relieve pain. During this period, the use of non-steroidal medication is forbidden.

Patients are prospectively evaluated basally and at 2, 6, and 12 months of follow-up using clinical subjective scores and objective parameters to determine clinical outcome (see 'Outcome measure' section). Patient satisfaction and adverse events will be also reported. All the clinical evaluations are performed by a medical staff not involved in the injective procedure, in order to keep the study double blinded. At the end of the study, the nature of the injected substance is revealed to the patients.

ELIGIBILITY:
Inclusion Criteria:

1. patients affected by mono-lateral symptomatic knee articular degenerative pathology with history of chronic (for at least 4 months) pain or swelling;
2. imaging findings of degenerative changes of the joint (osteoarthritis or chondropathy with Kellgren Lawrence Score from 0 to 3 at X-ray evaluation).

Exclusion Criteria:

* age > 80 years;
* Kellgren-Lawrence score at X-ray evaluation > 3;
* major axial deviation (varus >5° , valgus > 5°),
* systemic disorders such as diabetes, rheumatoid arthritis, haematological diseases (coagulopathy), severe cardiovascular diseases, infections, immunodepression;
* patients in therapy with anticoagulants or antiaggregants;
* use of NSAIDs in the 5 days before blood donation;
* patients with Hb values < 11 g/dl and platelet values < 150,000/mmc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2016-09-26 (Actual); Primary Completion 2017-09-26 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
IKDC (International knee documentation committee) score trend over time | basal (i.e. pre-treatment), 1 month, 2 months, 6 months and 12 months after treatment

SECONDARY OUTCOMES:
KOOS (Knee Outcome Osteoarthritis Score) trend over time | basal (i.e. pre-treatment), 1 month, 2 months, 6 months and 12 months after treatment
VAS (Visual Analogue Scale) for Pain trend over time | basal (i.e. pre-treatment), 1 month, 2 months, 6 months and 12 months after treatment
Tegner Score trend over time | basal (i.e. pre-treatment), 1 month, 2 months, 6 months and 12 months after treatment
Adverse events report during follow-up period | ba1 month, 2 months, 6 months and 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Berardo Di Matteo, MD, Study Chair — I Clinic, Rizzoli Orthopaedic Institute, Bologna, Italy; Alessandro Di Martino, MD, Study Chair — I Clinic, Rizzoli Orthopaedic Institute, Bologna, Italy; Francesco Tentoni, MD, Study Chair — I Clinic, Rizzoli Orthopaedic Institute, Bologna, Italy; Alice Roffi, BA, Study Chair — Rizzoli Orthopaedic Institute, Bologna, Italy; Elizaveta Kon, MD, Principal Investigator — I Clinic, Rizzoli Orthopaedic Institute, Bologna, Italy
Locations (1):
- Rizzoli Orthopaedic Institute, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Di Matteo B, Loibl M, Andriolo L, Filardo G, Zellner J, Koch M, Angele P. Biologic agents for anterior cruciate ligament healing: A systematic review. World J Orthop. 2016 Sep 18;7(9):592-603. doi: 10.5312/wjo.v7.i9.592. eCollection 2016 Sep 18. PMID 27672573
- [Background] van Drumpt RA, van der Weegen W, King W, Toler K, Macenski MM. Safety and Treatment Effectiveness of a Single Autologous Protein Solution Injection in Patients with Knee Osteoarthritis. Biores Open Access. 2016 Aug 1;5(1):261-8. doi: 10.1089/biores.2016.0014. eCollection 2016. PMID 27668131
- [Background] Mlynarek RA, Kuhn AW, Bedi A. Platelet-Rich Plasma (PRP) in Orthopedic Sports Medicine. Am J Orthop (Belle Mead NJ). 2016 Jul-Aug;45(5):290-326. PMID 27552452
- [Background] Sanchez M, Delgado D, Sanchez P, Muinos-Lopez E, Paiva B, Granero-Molto F, Prosper F, Pompei O, Perez JC, Azofra J, Padilla S, Fiz N. Combination of Intra-Articular and Intraosseous Injections of Platelet Rich Plasma for Severe Knee Osteoarthritis: A Pilot Study. Biomed Res Int. 2016;2016:4868613. doi: 10.1155/2016/4868613. Epub 2016 Jul 4. PMID 27462609
- [Background] Mariani E, Canella V, Cattini L, Kon E, Marcacci M, Di Matteo B, Pulsatelli L, Filardo G. Leukocyte-Rich Platelet-Rich Plasma Injections Do Not Up-Modulate Intra-Articular Pro-Inflammatory Cytokines in the Osteoarthritic Knee. PLoS One. 2016 Jun 3;11(6):e0156137. doi: 10.1371/journal.pone.0156137. eCollection 2016. PMID 27258008
- [Background] Sadabad HN, Behzadifar M, Arasteh F, Behzadifar M, Dehghan HR. Efficacy of Platelet-Rich Plasma versus Hyaluronic Acid for treatment of Knee Osteoarthritis: A systematic review and meta-analysis. Electron Physician. 2016 Mar 25;8(3):2115-22. doi: 10.19082/2115. eCollection 2016 Mar. PMID 27123220
- [Background] Yang J, Lu Y, Guo A. Platelet-rich plasma protects rat chondrocytes from interleukin-1beta-induced apoptosis. Mol Med Rep. 2016 Nov;14(5):4075-4082. doi: 10.3892/mmr.2016.5767. Epub 2016 Sep 23. PMID 27665780
- [Background] Yin WJ, Xu HT, Sheng JG, An ZQ, Guo SC, Xie XT, Zhang CQ. Advantages of Pure Platelet-Rich Plasma Compared with Leukocyte- and Platelet-Rich Plasma in Treating Rabbit Knee Osteoarthritis. Med Sci Monit. 2016 Apr 17;22:1280-90. doi: 10.12659/msm.898218. PMID 27086145
- [Background] Smyth NA, Haleem AM, Ross KA, Hannon CP, Murawski CD, Do HT, Kennedy JG. Platelet-Rich Plasma May Improve Osteochondral Donor Site Healing in a Rabbit Model. Cartilage. 2016 Jan;7(1):104-11. doi: 10.1177/1947603515599190. PMID 26958322
- [Background] Smith PA. Intra-articular Autologous Conditioned Plasma Injections Provide Safe and Efficacious Treatment for Knee Osteoarthritis: An FDA-Sanctioned, Randomized, Double-blind, Placebo-controlled Clinical Trial. Am J Sports Med. 2016 Apr;44(4):884-91. doi: 10.1177/0363546515624678. Epub 2016 Feb 1. PMID 26831629
- [Derived] Di Martino A, Boffa A, Andriolo L, Romandini I, Altamura SA, Cenacchi A, Roverini V, Zaffagnini S, Filardo G. Leukocyte-Rich versus Leukocyte-Poor Platelet-Rich Plasma for the Treatment of Knee Osteoarthritis: A Double-Blind Randomized Trial. Am J Sports Med. 2022 Mar;50(3):609-617. doi: 10.1177/03635465211064303. Epub 2022 Feb 1. PMID 35103547